CLINICAL TRIAL: NCT04572698
Title: To Compare the Efficacy and Safety of Recombinant Human Vascular Endothelial Growth Factor Receptor Antibody Fusion Protein Eye Injection（LY09004） and Eylea in the Treatment of Wet Age-related Macular Degeneration（wAMD）: a Randomized, Double-blind, Parallel Controlled, Multicenter Clinical Trial
Brief Title: A Study to Compare LY09004 and Eylea in the Treatment of Wet Age-related Macular Degeneration（wAMD）
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Luye Pharma Group Ltd. (Industry)
Collaborators: Shan Dong Boan Biotechnology Co., Ltd(Co-sponsor) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LY09004/CT-CHN-302
Record Dates: First submitted 2020-09-21; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Age Related Macular Degeneration
Keywords: w-AMD; LY09004; EYLEA; efficacy; safety
MeSH Terms: conditions — Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY09004 (Experimental): LY09004 injection by intraocular injection on Day1, Day29, Day57,Day113, Day169, Day225, Day281 and Day337.
  Interventions: Drug: LY09004
- EYLEA (Active Comparator): EYLEA injection by intraocular injection on Day1, Day29, Day57,Day113, Day169, Day225, Day281 and Day337.
  Interventions: Drug: Eylea

INTERVENTIONS:
Drug: LY09004 — LY09004 injection by intraocular injection on Day1, Day29, Day57,Day113, Day169, Day225, Day281 and Day337.
  Other Names: Recombinant Human Vascular Endothelial Growth Factor Receptor Antibody Fusion Protein Eye Injection
  Arms: LY09004
Drug: Eylea — EYLEA injection by intraocular injection on Day1, Day29, Day57,Day113, Day169, Day225, Day281 and Day337.
  Arms: EYLEA

SUMMARY:
A randomized, double-blind, parallel controlled, multicenter clinical trial to compare the efficacy and safety of LY09004 and EYLEA in the Treatment of Wet Age-related Macular Degeneration（wAMD)

DETAILED DESCRIPTION:
This is a randomized, double-blind, parallel controlled, multicenter clinical trial.

The primary objective is to assess the efficacy similarity of LY09004 and EYLEA in the treatment of w-AMD.

The secondary objective is to assess the safety similarity of LY09004 and EYLEA in the treatment of w-AMD.

ELIGIBILITY:
Inclusion Criteria:

1. The patient or their legal representatives must give the written informed consent form voluntarily;
2. Aged ≥ 50 years, male or female;
3. Patients confirmed diagnosis of w-AMD, currently have active lesions, which are defined any of the following in the macular area: ① intraretinal fluid; ② intraretinal lipid exudation; ③ subretinal fluid; ④ subretinal hemorrhage; ⑤ retinal pigment epithelium detachment;
4. The total area of all types of lesions in the study eye ≤ 30mm2 (the area of 12 optic discs);
5. The BCVA between 73-24 letters (including boundary values) in the study eye is inclusive using the ETDRS, which is equivalent to 20/40 to 20/320 of Snellen；
6. Non-study eye use ETDRS testing to detect BCVA ≥19 letters，which is equivalent to 20/400 of Snellen;
7. At hte time of screening, childbearing-age (such as women who have not undergone surgical sterilization or have been postmenopausal less than one year) have a negative blood pregnancy test result. Childbearing-age male and female agree to take effective contraceptive measures throughout the study period and for at least 3 months after medication.

Exclusion Criteria:

1. Any opacity of refractive media or non-dilated pupils in the study eye interference with visual acuity detection and the evaluation of anterior segment and fundus;
2. Study eye retinal hemorrhage ≥ 4 optic disc area;
3. Central fovea of the study eye affected by geographic atrophy, scars or fibrosis, dense subfoveal exudation, and macula center affected by retinal pigment epithelium (RPE) tear;
4. Any concurrent conditions in the study eye that affects central vision (such as diabetic retinopathy, retinal vein occlusion, uveitis, vascular streaks, pathological myopia, retinal detachment, macular hole, epimacular membrane, toxoplasmosis , Optic nerve disease, polypoid choroidal vascular disease (PCV), etc.);
5. Any history of the following ophthalmic surgery in the study eye: vitrectomy, anti-glaucoma surgery, macular transposition;
6. Any evidence of external eye surgery within 1 month or cataract surgery within 3 months before screening in the study eye;
7. Any the following treatment in the study eye within 3 months before screening: Verteporfin photodynamic therapy (PDT), macular laser photocoagulation, transpupillary thermotherapy (TTT), and other operations for the treatment of AMD;
8. Aphakia (excluding intraocular lens) or posterior lens capsule rupture (except for YAG laser posterior capsulotomy after intraocular lens implantation more than 1 month from screening) in the study;
9. Afferent pupil defect (APD) in the study eye;
10. Patients have received anti-VEGF(vascular endothelial growth factor ) treatment within 6 months before screening, such as ranibizumab, bevacizumab, conbercept, etc in any eye or the whole body;
11. Use of intraocular or systemic corticosteroids within 3 months before screening, or use of periocular corticosteroids within 1 month;
12. Any active intraocular or periocular infection (for example: blepharitis, infectious conjunctivitis, keratitis) in either eye;
13. Any history of glaucoma;
14. Any evidence of pseudocapsular exfoliation syndrome in either eye;
15. A history of vitreous hemorrhage within 3 months before screening in either eye;
16. Any systemic drug (currently in use or may need to use) could cause lens toxicity or retinal toxicity, such as desferrioxamine, chloroquine/hydroxychloroquine, tamoxifen, phenothiazine, ethambutol, etc.;
17. History of allergy to the therapeutic or diagnostic drugs used in the research protocol, including allergies to the test articles;
18. Diabetic subjects with diabetic retinopathy or glycosylated hemoglobin> 9%;
19. Any history of surgery within 1 month before screening, and/or any currently unhealed wounds, ulcers, fractures, etc.;
20. Any infectious disease requiring systemic treatment (oral, intramuscular or intravenous) during screening;
21. History of a medical condition, including myocardial infarction, unstable angina pectoris, coronary revascularization, cerebrovascular accidents (including TIA), other thromboembolic diseases (such as thromboembolic angiitis, pulmonary embolism, deep vein thrombosis, portal vein thrombosis, etc.), New York Heart Association (NYHA) grade ≥ Grade II cardiac insufficiency, severely unstable ventricular arrhythmia within 6 months before screening;
22. History of diffuse intravascular coagulation and obvious bleeding tendency (such as hemoptysis, hematemesis, severe purpura, etc.) within 3 months before screening, or use of anticoagulant and antiplatelet therapy other than aspirin/NSAIDs within 14 days before screening;
23. Subjects with systemic immune diseases;
24. Poorly-controlled blood pressure (defined as: after receiving antihypertensive drugs, the subject's systolic value ≥160 mmHg or diastolic value ≥100 mmHg at seat);
25. Any uncontrollable clinical disease (such as serious mental, respiratory and other system diseases and malignant tumors);
26. Abnormal liver and kidney function (ALT, AST≥2.5 times the upper limit of normal; total bilirubin≥1.5 times the upper limit of normal; Crea, urea/urea nitrogen≥1.2 times the upper limit of normal);
27. Abnormal blood coagulation function (prothrombin time> upper limit of normal value 3 seconds or activated partial thromboplastin time> upper limit of normal value 10 seconds);
28. Positive Hepatitis B surface antigen (HBsAg), and peripheral blood hepatitis B virus deoxyribonucleic acid (HBV DNA) titer test ≥ 1 × 103 copies/mL; Under the condition of positive HBsAg with peripheral blood HBV DNA titer test <1x 103 copies/mL, if the investigator judges that chronic hepatitis B is stable and will not increase the risk of the subject, the subject is eligible for selection;
29. Positive Hepatitis C virus (HCV) antibody, Treponema pallidum antibody, and human immunodeficiency virus (HIV) antibody;
30. Nursing (lactating) women;
31. Participation in clinical trials of any drug (excluding vitamins and minerals) within 3 months before screening;
32. Others need to be excluded according to the judgement of the investigator.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
BCVA（best corrected visual acuity ） | week 24
  Assess the BCVA change similarity from baseline of LY09004 and EYLEA

SECONDARY OUTCOMES:
BCVA | week 4, week 8, week 12, week 16, week 20, week 28, week 32, week 36, week 40, week 44, week 48, week 52
  Assess the BCVA change similarity from baseline of LY09004 and EYLEA
Letter | week 24, week 52
  Proportion of subjects with 5 / 10 / 15 letters more than baseline in study eye
Central television omentum thickness | week 24, week 52
  Changes of central television omentum thickness from baseline in study eyes
CNV(Choroidal neovascularization) leakage area | week 24, week 52
  Changes of CNV leakage area of study eye compared with baseline

OTHER OUTCOMES:
AE(adverse event) | week 52
  Number of patients with treatment related adverse events assessed by change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Youxin Chen, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No